CLINICAL TRIAL: NCT04878666
Title: Prospektive Erfassung Der Lebensqualität Bei Patientinnen Mit Lokal Rezidiviertem Mammakarzinom Und Hyperthermer Radiotherapie (UKT HT03.1)
Brief Title: Prospective Assessment of Quality of Life in Patients With Locally Recurrent Breast Cancer and Hyperthermic Radiotherapy
Acronym: UKT HT03_1
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: UKT HT03_1
Record Dates: First submitted 2021-03-08; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: Hyperthermic Radiotherapy; Quality of Life; locally recurrent Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective assessment of Quality of Life in patients with locally recurrent breast cancer after close R0, R1 or R2 resection or local inoperability and hyperthermic radiotherapy.

DETAILED DESCRIPTION:
This prospective monocentric trial evaluates the health-related Quality of Life in patients with local recurrence of Breast cancer after close R0, R1 or R2 resection or local inoperability during and after radiotherapy in combination with hyperthermia of the chest wall. The Health-related Quality of Life and the intensity of fatigue will be documented by the EORTC QLQ-C30, EORTC QLQ - BR 23, FACT - B + 4 and FACIT - Fatigue Questionnaires at the end of the hypertermic radiotherapy and during follow-up after 3 and 12 month and then annually up to year 5.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed local recurrence of breast cancer after close resection (≤1mm Resection margin), R1 or R2 resection respectively inoperable recurrence of the chest wall
* age ≥18 Jahre
* ECOG PS 0-2
* Estimated life expectancy more than 2 years
* Informed consent

Exclusion Criteria:

* Extensive distant metastases that have an estimated life expectancy of <2a
* Heart disease: severe heart failure (NHYA III / IV), coronary heart disease, state after Myocardial infarction within the last 6 months), AV block III °
* Cardiac pacemaker
* Second malignancy (except cervical carcinomas in situ, local controlled basaliomas, superficial bladder carcinomas (Ta, Tis, T1) or other carcinomas that have lasted more than 5 years behind and have been treated curatively)
* Pregnancy or breastfeeding
* Implanted port on the side to be treated in the Hyperthermia field (located contralateral is not an exclusion criteria)
* Subclavian vein thrombosis less than <6 months behind
* Other circumstances that preclude hyperthermia
* Circumstances that conflict with regular follow-up care
* Transplanted organs
* Other implants of the ipsilateral chest wall

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a histologically confirmed local recurrence of breast cancer after close R0, R1 or R2 resection respectively inoperable recurrence of the chest wall with or without a previous irradiation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the health-related Quality of Life (QoL) during and after hyperthermic radiotherapy. QoL will be measured by the EORTC QLQ BR 23 | During hyperthermic radiotherapy up to five years of follow-up.
  Assessment of the health-related QoL in patients who receive a surface hyperthermia in parallel with a radiotherapy of the chest wall as part of a multimodal therapy. This endpoint will be evaluated by the -BR 23 subscale (4 functional subscales, 4 symptom subscales.All subscales have a point value range from 0 to 100 points. A higher score represents better function and a higher quality of life. With symptom subscales, however, a higher score represents a higher level of symptoms or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Heinrich, MD, Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Department of Radiation Oncology, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No